CLINICAL TRIAL: NCT04903860
Title: Comparison of the Use of Conventional Ancillary Reaming and Single-use Ancillary Reaming Material in Total Hip Replacement
Acronym: LUUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Groupe Lépine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2021 ERIVAN; 2021-A00363-38 (Other: 2021-A00363-38)
Record Dates: First submitted 2021-05-12; First posted 2021-05-27 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Total Hip Replacement; Coxarthrosis
Keywords: Prospective; Randomized study; Medico-economic; Sterilization; Single use reamer; Ancillary
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single use reamers (Active Comparator): Total hip replacement with the use of disposable reamers
  Interventions: Device: total hip replacement with single use ancillary
- conventional ancillary (Active Comparator): Total hip replacement with the use of conventional reamers
  Interventions: Device: total hip replacement with conventional ancillary

INTERVENTIONS:
Device: total hip replacement with single use ancillary — Comparison of the use of conventional ancillary reaming and single-use ancillary reaming material in total hip replacement
  Arms: Single use reamers
Device: total hip replacement with conventional ancillary — Comparison of the use of conventional ancillary reaming and single-use ancillary reaming material in total hip replacement
  Arms: conventional ancillary

SUMMARY:
The main objective of the study is to compare the use of single-use ancillary reaming material during total hip replacement and conventional reusable ancillary reaming material.

The assessment will focus on the medico-economic differences found in this prospective randomized study

DETAILED DESCRIPTION:
In orthopaedics, the ancillary equipment is a generic term that includes all the instruments necessary for hip replacement surgery. The surgeon remains very dependent on these boxes of instruments, including rasps, reamers and trial implants (stems and trial heads), which are required in THR. Each instrument set is generally packaged in 2 or 3 boxes and each surgeon has a limited number of instrument sets at his disposal per operating day. Each ancillary device has a purchase cost, a maintenance cost (paid by the laboratories or distributors) and a sterilization cost, (paid by the health care institutions).

Single-use reamers are instruments that are used on a single patient and then discarded. Performance and safety of use are optimized by providing a sterile and new product for each use.

Therefore, it seems judicious to compare the medico-economic differences between the use of single-use reamers versus reusable reamers within a classic ancillary.

This study will compare the costs incurred, the waste produced, the operating time, the satisfaction of the surgeon after the use of single-use reamers during total hip replacement, versus conventional re-sterilizable ancillary and verify the equivalence, three months after surgery, of clinical and radiological results.

ELIGIBILITY:
Inclusion Criteria:

* - Patient, male or female, over 18 years of age, eligible for a first-line total hip replacement for isolated coxarthrosis
* Patient registered to the national health system
* Patient able to understand information about the protocol and answer to questionnaire

Exclusion Criteria:

* Pregnant, breastfeeding or potentially pregnant woman
* Major disability
* History of hip replacement surgery
* Any surgical and/or anesthetic contraindication, or any condition deemed by the investigator to be incompatible with the research.
* Morbid obesity as defined by body mass index (BMI) >40 kg.m-2
* History of recent infection at the surgical site
* Surgical contraindication
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Overall cost of surgery | At 3 months
  Direct medical costing in both groups:
  * Sterilization costs,
  * Inventory management costs,
  * Material costs,
  * Waste management costs,
  * Operating room costs based on room occupancy times.

SECONDARY OUTCOMES:
Surgical time | intraoperative
  Calculated from the beginning of the skin incision to closure and recorded on the anesthesia sheet
Modified Merle d'Aubigné and Postel Method score | Pré-opérative examination / At 3 months
  The patients were evaluated by the Modified Merle d'Aubigné and Postel Method, which evaluates pain, gait and mobility, on a scale of 1 to 6 for each item, where 1 indicates the worst and 6, the best state of the patient. The total minimum score reached is 3, and the maximum is 18.
Harris Hip Score | Pré-opérative examination / At 3 months
  This instrument has 10 items in 3 sections describing pain, function, range of motion, and deformity. The first section is questionnaire-based, answered by the patient, and includes impairments and activities. The second and third sections are administered by the therapist or physician, and include leg length measurement and range of motion (ROM) measures of the hip (flexion, abduction, external rotation and adduction). Each item has a unique numerical scale that corresponds to descriptive response options. The highest possible score is 100, with a higher score indicating less dysfunction.
Charnley classification and Devane score | Pré-opérative examination / At 3 months
  Devane score: The purpose of this score is to specify the patient's activity level preoperatively. Initially established by Devane, it allows a classification of each patient in 5 categories from sedentary to athletic Charnley score: This is a commonly used score designed to assess the patient's overall disability in relation to gait function. It was published by Charnley and distinguishes patients into 3 categories
WOMAC score | Pré-opérative examination / At 3 months
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of hip, including five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68).
HOOS score | Pré-opérative examination / At 3 months
  The hip disability and osteoarthritis outcome score (HOOS) is a questionnaire intended to be used to assess the patient's opinion about their hip and associated problems and to evaluate symptoms and functional limitations related to the hip during a therapeutic process. To interpret the score, the outcome measure is transformed in a worst to best scale from 0 to 100, with 100 indicating no symptoms and 0 indicating extreme symptoms.
Pain evaluation | Pré-opérative examination / At 3 months
  The visual similar scale is auto completed. For the intensity of pain, the scale varies between "no pain" (the score of 0) and "most painful" (the score of 10).
Operator satisfaction | through surgical intervention an average of 1 day
  Operator satisfaction score (numerical scale from 0 (not satisfied) to 10 (very satisfied)) of the material during the surgical procedure
Radiological analysis | At 3 months
  realization of standard radiographs of the pelvis from the front, hip from the front and from the side. Analysis of the acetabulum according to Charnley and search for the presence of granulometry, migration or acetabular osteolysis. Measurement of the femoral and acetabular offset and height of the center of rotation
Complications | At 3 months
  Analysis of possible intraoperative and postoperative complications and their costs: loosening, infection, dislocation, wear and implant fracture

CONTACTS AND LOCATIONS:
Overall Officials: Roger ERIVAN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Erivan R, Bourzat N, Mulliez A, Mougues C, Descamps S, Boisgard S, Villatte G. Single-use versus reusable ancillaries for dual mobility cup in total hip replacement. A prospective randomized short-term safety and feasibility comparison. Orthop Traumatol Surg Res. 2023 Nov;109(7):103658. doi: 10.1016/j.otsr.2023.103658. Epub 2023 Jul 13. PMID 37451339